CLINICAL TRIAL: NCT01706237
Title: Evaluation Of Visual Outcomes And Contrast Sensitivity After Myopic Wavefront-Optimized Lasik With Nexisvision Shield Or Bandage Contact Lens
Brief Title: Visual Outcomes And Contrast Sensitivity After Myopic Wavefront-Optimized Lasik With Nexisvision Shield Or Bandage Contact Lens
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Nexis Vision was unable to provide the shields to continue with the study.
Sponsor: Durrie Vision (Other)
Collaborators: Nexisvision (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NVS-SOVR-001
Record Dates: First submitted 2012-10-11; First posted 2012-10-15 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Myopia
Keywords: Myopia; LASIK
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Shield (Experimental): A shield (similar to a contact lens) is placed on the eye after myopic LASIK procedure.
  Interventions: Device: Nexisvision shield

INTERVENTIONS:
Device: Nexisvision shield — A shield is placed on the eye after LASIK. The shield is similar to a contact lens.

SUMMARY:
Evaluate visual outcomes and contrast sensitivity for subjects undergoing bilateral myopic LASIK with a Nexisvision Shield or bandage contact lens placed postoperatively. Early speed of visual recovery results indicate that the visual recovery in the first 4 hours after the LASIK procedure show the most variability. A patient's ability to drive after their LASIK procedure would potentially alleviate a challenge that patients often face in taking additional time off work or simply finding a ride to there LASIK procedure.

DETAILED DESCRIPTION:
Laser in situ keratomileusis (LASIK) surgery has been performed worldwide since 1990. Historically, LASIK has been reported to decrease contrast sensitivity post operatively and patients have been advised to take the day off of work and potentially the day after LASIK. More recently, utilizing advanced laser technology for optimized corneal ablation and creation of the flap has the potential for improved LASIK surgery results and improved recovery time. Visual recovery and management of immediate post operative visual acuity is important for patient satisfaction.

ELIGIBILITY:
INCLUSION CRITERIA:

* Male or female in good general health, 18 years of age or older at the time of the pre-operative examination
* Patient must be able to read, comprehend and willing to give HIPPA and informed consent
* Patient is planning to undergo a bilateral LASIK procedure
* Both eyes must have a manifest refractive error from -1.00 D to -7.00 spherical equivalent with less than or equal to 3.00D of refractive astigmatism as expressed in spectacle minus cylinder form
* Both eyes must have a BSCVA of 20/20 or better
* Both eyes must demonstrate refractive stability confirmed by clinical records, previous glasses, or investigator's discretion.
* Patient must be willing to comply with study dosing and complete the entire course of the study.

EXCLUSION CRITERIA:

* A patient with evidence of keratoconus, corneal irregularity, or abnormal videokeratography in either eye
* A patient seeking monovision
* A patient with a known hypersensitivity to any of the components of the procedural or post-LASIK medications
* A patient requiring the use of any ocular drop(s) and/or medication(s) in either eye during the study period with the exception of ocular drops and/or medications provided by the investigator
* A patient having any surgical procedure within a week preceding the scheduled LASIK surgery
* A patient with any UNCONTROLLED systemic disease (i.e., a potential patient in whom therapy for a systemic disease is not yet stabilized )
* A patient with a history of prior intraocular or corneal surgery (including cataract extraction), active ophthalmic disease or abnormality (including, but not limited to, blepharitis, recurrent corneal erosion, dry eye syndrome, neovascularization > 1mm from limbus), clinically significant lens opacity, clinical evidence of trauma (including scarring), or evidence of glaucoma or propensity for narrow angle glaucoma in either eye
* A patient with a significant history or current evidence of a medical, psychological or other disorder that, in the investigator's opinion, may increase the risk associated with study participation or may interfere with the interpretation of study results
* A patient with a history of any of the following medical conditions, or any other condition that could affect wound healing: uncontrolled diabetes, collagen vascular disease, autoimmune disease, immunodeficiency diseases, ocular herpes zoster or simplex, endocrine disorders (including, but not limited to unstable thyroid disorders and diabetes), lupus, and rheumatoid arthritis
* Current participation or participation within 30 days prior to the start of this study in a drug or other investigational research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-05; Primary Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Visual Acuity over time | Immediate, 30 minutes, 1 hour, 2 hour, and 4 hours
  Progress of the change in visual acuity will be measured at specific time intervals directly after LASIK surgery.
Contrast Sensitivity | Immediate, 30 minutes, 1 hour, 2 hour, and 4 hours
  Change in contrast sensitivity compared to baseline will be documented at specific time intervals beginning immediately after LASIK surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Durrie, MD, Principal Investigator — Durrie Vision; Stephen G. Slade, MD, Principal Investigator — Slade & Baker Vision